CLINICAL TRIAL: NCT01940510
Title: An Open-Label, Three-Period, Fixed Sequence Study to Investigate the Effect of Multiple Oral Doses of Rifampin, a Potent Cytochrome P450 3A Inducer, on the Single Dose Pharmacokinetics of RO5424802 in Healthy Subjects
Brief Title: A Study of the Effect of Multiple Doses of Rifampin on the Single Dose Pharmacokinetics of RO5424802
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NP29042
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — alectinib; Rifampin

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Drug: RO5424802; Drug: rifampin

INTERVENTIONS:
Drug: RO5424802 — Single dose without (Day 1) and with (Day 17) co-administration of rifampin
Drug: rifampin — Multiple doses Days 8-16 and Days 17-20

SUMMARY:
This single center, open-label, 3-period, fixed-sequence study will evaluate the effect of multiple oral doses of rifampin on the pharmacokinetics of a single oral dose of RO5424802 in healthy volunteers. Subjects will receive a single dose of RO5424802 on Days 1 and 17 and rifampin daily from Days 8 to Day 20.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 to 55 years of age inclusive. Healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, and a complete physical examination
* Body mass index (BMI) between 18 to 32 kg/m2 inclusive
* Nonsmoking subjects and former smoking subjects (who have not smoked for the past six months before first dosing)
* Female subjects must be surgically sterile or postmenopausal for the past year
* Male subjects and their partners of childbearing potential must be willing to use two effective methods of contraception, one of which must be a barrier method (e.g., condom) during the study and for 90 days after the last drug administration

Exclusion Criteria:

* Women of childbearing potential, pregnant or lactating women, or males with female partners who are pregnant or lactating
* Positive urine test for drugs of abuse, alcohol, or cotinine test at screening or prior to admission to the study unit
* Suspicion of regular consumption of drug(s) of abuse including marijuana
* Current smokers or subjects who have discontinued smoking less than six months prior to first dosing
* History (within three months of Screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol). Alcohol consumption will be prohibited 72 hours prior to entry in the clinical site center and throughout the entire study (including the washout period) until discharge
* Positive for hepatitis B, hepatitis C, or HIV infection
* Participation in an investigational drug or device study within 45 days or 5 half-lives (whichever time period is longer) or 6 months for biologic therapies prior to first dosing
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, absorption, distribution, metabolism or excretion of study medication, or that would, in the opinion of the PI, pose an unacceptable risk to the subject in this study
* History of hypersensitivity to any of the additives in the RO5424802 formulation (lactose monohydrate, microcrystalline cellulose, sodium starch glycolate, hydroxypropyl cellulose, sodium lauryl sulphate, magnesium stearate)
* Any history of hypersensitivity to or contraindication to the use of rifampin or other rifamycins or history of severe drug-related allergic reactions or hepatoxicity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Study: Alectinib + Rifampin: There were 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 16), and Period 3 (Days 17 to 21). Participants following an overnight fast of at least 10 hours ate a standard meal in 30 minutes or less and 30 minutes after start of the meal received alectinib (RO5424802) 600 milligram (mg) capsules (four 150 mg capsules) orally alone on Day 1 (Period 1), with rifampin (600 mg capsules [two 300 mg capsules] orally) on Day 17 (Period 3), and rifampin alone was administered from Days 8 through 16 (Period 2) and from Days 18 through 20 (Period 3).
Period: Overall Study
Arm/Group | Whole Study: Alectinib + Rifampin
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of the study treatment and had at least 1 postdose safety assessment.
Groups:
- Whole Study: Alectinib + Rifampin: There were 3 dosing periods in the study: Period 1 (Days 1 to 7), Period 2 (Days 8 to 16), and Period 3 (Days 17 to 21). Participants following an overnight fast of at least 10 hours ate a standard meal in 30 minutes or less and 30 minutes after start of the meal received alectinib 600 mg capsules orally alone on Day 1 (Period 1), with rifampin (600 mg capsules orally) on Day 17 (Period 3), and rifampin alone was administered from Days 8 through 16 (Period 2) and from Days 18 through 20 (Period 3).
Arm/Group | Whole Study: Alectinib + Rifampin
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.43)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Alectinib
Description: AUC(0-inf) is the area under the alectinib plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of a drug over time. AUC(0-inf) is presented in nanogram times (*) hour per milliliter (ng*hour/mL).
Time Frame: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours post alectinib-dose in each intervention period
Population: The Pharmacokinetic (PK) analysis set included all participants who received both scheduled doses of alectinib (on Day 1 and Day 17), and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Groups:
- Treatment Period 1: Alectinib: Participants following an overnight fast of at least 10 hours ate a standard meal in 30 minutes or less and 30 minutes after start of the meal received alectinib 600 mg capsules orally on Day 1 of treatment period 1.
- Treatment Period 3: Alectinib + Rifampin: Participants following an overnight fast of at least 10 hours ate a standard meal in 30 minutes or less and 30 minutes after start of the meal received alectinib 600 mg capsules orally on Day 1 of treatment period 3 (Day 17). Participants following an overnight fast of at least 10 hours received rifampin 600 mg capsules orally once daily from Day 18 through 20. On Day 17, rifampin was coadministered with alectinib, 30 minutes after start of the standard meal.
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ng*hour/mL | 3990 (1550) | 1020 (240)
Statistical Analysis 1: Comparison: Treatment Period 1: Alectinib vs Treatment Period 3: Alectinib + Rifampin; Analysis of variance (ANOVA) was applied to the log-transformed PK parameters, and then back transformed to provide geometric least square mean ratios (Period 3/Period 1) and confidence intervals; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 26.8, 90% CI 2-sided [23.8 to 30.1] — The reported values are percentages of geometric least square mean ratio

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Alectinib
Description: Cmax is the maximum observed alectinib plasma concentration, presented in nanogram per milliliter (ng/mL).
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ng/mL | 212 (78.3) | 101 (30.9)
Statistical Analysis 1: Comparison: Treatment Period 1: Alectinib vs Treatment Period 3: Alectinib + Rifampin; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 48.6, 90% CI 2-sided [43.5 to 54.3] — ANOVA was applied to the log-transformed PK parameters, and then back transformed to provide geometric least square mean ratios (Period 3/Period 1) and confidence intervals. The reported values are percentages of geometric least square mean ratio

3. Secondary Outcome: AUC(0-inf) of RO5468924
Description: AUC(0-inf) is the area under the RO5468924 (the major pharmacologically active metabolite of alectinib) plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of the drug over time. AUC(0-inf) is presented in ng*hour/mL.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ng*hour/mL | 2250 (904) | 3970 (1600)
Statistical Analysis 1: Comparison: Treatment Period 1: Alectinib vs Treatment Period 3: Alectinib + Rifampin; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 179, 90% CI 2-sided [158 to 202] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Cmax of RO5468924
Description: Cmax is the maximum observed RO5468924 (the major pharmacologically active metabolite of alectinib) plasma concentration, presented in ng/mL.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ng/mL | 90.5 (43.7) | 194 (97.0)
Statistical Analysis 1: Comparison: Treatment Period 1: Alectinib vs Treatment Period 3: Alectinib + Rifampin; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 220, 90% CI 2-sided [190 to 255] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for AUC(0-inf)
Description: AUC(0-inf) is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib) over time. The molecular weight adjusted M/P ratio (RO5468924/alectinib) for AUC(0-inf) is presented.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ratio | 0.59 (0.05) | 3.96 (0.67)

6. Secondary Outcome: Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for Cmax
Description: Cmax is the maximum observed plasma concentration of the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib). The molecular weight adjusted M/P ratio (RO5468924/alectinib) for Cmax is presented.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ratio | 0.42 (0.07) | 1.92 (0.32)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) of Alectinib and RO5468924
Description: AUC(0-last) is the area under the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib) plasma concentration time-curve from time zero to the last measured concentration. AUC is a measure of the plasma concentration of a drug over time. AUC(0-last) is presented in ng*hour/mL.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
ng*hour/mL
  Alectinib | 3860 (1500) | 976 (234)
  RO5468924 | 2140 (876) | 3850 (1570)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alectinib and RO5468924
Description: The Tmax is the time from alectinib administration to reach Cmax for alectinib and RO5468924 (the major pharmacologically active metabolite of alectinib).
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
hours
  Alectinib | 6.00 [4.00 to 12.00] | 4.00 [4.00 to 8.00]
  RO5468924 | 8.00 [6.00 to 12.00] | 6.00 [6.00 to 8.00]

9. Secondary Outcome: Plasma Terminal Half-Life (t1/2) of Alectinib and RO5468924
Description: Plasma terminal half-life is the time measured during drug elimination phase for the plasma drug concentration to decrease by one half. RO5468924 is the major pharmacologically active metabolite of alectinib.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
hours
  Alectinib | 19.2 (4.41) | 11.0 (5.65)
  RO5468924 | 24.0 (3.48) | 23.0 (11.1)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) of Alectinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
liters/hour | 179 (89.1) | 627 (170)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Alectinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction of drug absorbed.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
liters | 4710 (1890) | 9960 (5880)

12. Secondary Outcome: Total Molar Concentration of Alectinib and RO5468924 as Derived by AUC(0-inf)
Description: AUC(0-inf) is the area under the alectinib + RO5468924 (major pharmacologically active metabolite of alectinib) molar plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the molar plasma concentration of the alectinib + RO5468924 over time. AUC(0-inf) is presented in nanomoles times (*) hour per liter (nmol*hour/L).
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol*hour/L
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
nmol*hour/L | 13200 (4670) | 10800 (3910)

13. Secondary Outcome: Total Molar Concentration of Alectinib and RO5468924 as Derived by Cmax
Description: Cmax is the maximum observed molar plasma concentration for alectinib + RO5468924 (major pharmacologically active metabolite of alectinib). Cmax is presented in nanomoles per liter (nmol/L).
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 3: Alectinib + Rifampin
Number analyzed (Participants) | 24 | 24
nmol/L | 614 (231) | 594 (251)

ADVERSE EVENTS:
Time Frame: Day 1 through follow-up (up to 31 days)
Description: Safety analysis set. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment-emergent AE (TEAE) was defined as an AE that began or worsened in severity on or after the first dose of the study drug.
Groups:
- Treatment Period 2: Rifampin: Participants following an overnight fast of at least 10 hours received rifampin 600 mg capsules orally once daily from Day 8 through 16.
Arm/Group | Treatment Period 1: Alectinib | Treatment Period 2: Rifampin | Treatment Period 3: Alectinib + Rifampin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 16/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: Alectinib (N=24) | Treatment Period 2: Rifampin (N=24) | Treatment Period 3: Alectinib + Rifampin (N=24)
Chromaturia (Renal and urinary disorders) | 0 | 14 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.